CLINICAL TRIAL: NCT00998205
Title: Early Diagnosis of Diastolic Dysfunction and Reliability of Dobutamine Stress Echo (DSE) in Detecting Stress Diastolic Dysfunction
Brief Title: Early Diagnosis of Diastolic Dysfunction and Reliability of DSE in Detecting Stress Diastolic Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Kansas City Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1115797
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Diastolic Dysfunction
MeSH Terms: interventions — Dobutamine; Atropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dobutamine stress echo (DSE) (Other): Dobutamine intravenous infusion would be undertaken starting at 10 micrograms/kg per minute in three minute intervals increased to 20, 30, 40 or 50 micrograms/kg per minute or to a peak heart rate response of at least 85% age predicted maximum heart rate. If at the end of the Dobutamine protocol, there is inadequate heart rate response, intravenous atropine boluses of 0.5 milligrams (maximum 1.0 mg) would be used as needed to achieve a heart rate of at least 85% of age predicted maximum heart rate.
  Interventions: Drug: Dobutamine stress echo (DSE); Drug: Atropine bolus

INTERVENTIONS:
Drug: Dobutamine stress echo (DSE) — Dobutamine intravenous infusion would be undertaken starting at 10 micro-grams/kg per minute in three minute intervals increased to 20, 30, 40 or 50 micro-grams/kg per minute or to a peak heart rate response of at least 85% age predicted maximum heart rate.
  Other Names: Dobutamine hydrochloride
Drug: Atropine bolus — If at the end of the Dobutamine protocol, there is inadequate heart rate response, intravenous atropine boluses of 0.5 milligrams (maximum 1.0 mg) would be used as needed to achieve a heart rate of at least 85% of age predicted maximum heart rate.
  Other Names: Atropine sulfate

SUMMARY:
The heart becoming "stiff" due to increased fibrous tissue or decreased elasticity of the heart tissue is one of the earliest changes caused by heart failure. These changes can be detected by simple non-invasive echocardiogram techniques. However, these techniques usually detect the increased "stiffness" of the heart only after it has progressed to a significant extent. The investigators hypothesize that if they stress the heart using a Dobutamine infusion and measure the filling pressure using echocardiogram, it will provide them with tools to identify these changes earlier.

DETAILED DESCRIPTION:
The heart becoming "stiff" due to increased fibrous tissue or decreased elasticity of the heart tissue is one of the earliest changes caused by heart failure. These changes can be detected by simple non-invasive echocardiogram techniques. However, these techniques usually detect the increased "stiffness" of the heart only after it has progressed to a significant extent. The investigators hypothesize that if they stress the heart using a Dobutamine infusion and measure the filling pressure using echocardiogram, it will provide them with tools to identify these changes earlier.

The investigators are planning to include people have normal heart function. It is standard procedure to measure cardiac pressure during catheterization. Simultaneously, the investigators will infuse Dobutamine (standard drug used for chemical stress testing, DSE). This drug increases the heart rate and mimics exercise in normal humans who are unable to exercise for various reasons. The investigators would continue to monitor the pressure inside the heart as they infuse Dobutamine and see of there is an increase in filling pressure. The investigators will correlate the invasive pressures with their echo derived measurements.

The investigators plan to include 25 veterans in this study. For each individual the study would increase the amount of time they will spend in the Catheterization Lab from 30 to 120 minutes. The entire procedure will be monitored by Advanced Cardiac Life Support (ACLS) certified nurses and doctors.

ELIGIBILITY:
Inclusion Criteria:

* Prospectively enroll 25 veterans age range from 18 to 65 who are found to have normal left ventricular (LV) systolic function and no significant coronary artery disease by cardiac catheterization.
* Subjects identified during routine cardiac testing to have significant diastolic dysfunction may also be enrolled to rule out coronary disease and study DSE -invasive pressure correlations.

Exclusion criteria:

* Patients with LV systolic dysfunction, severe coronary lesions (> 50%), uncontrolled hypertension (BP > 160/100) and significant pulmonary hypertension (PASP > 50 mmHg) would be excluded.
* Subject will not be included if they have a significant rhythm abnormality, frequent premature ventricular complexes, atrial fibrillation and technical reasons in the catheterization laboratory which preclude the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anand Chockalingam, MD, Principal Investigator — University of Missouri/Harry S Truman VA Hospital
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Dobutamine Stress Echo (DSE): Dobutamine intravenous infusion starting at 10 micrograms/kg per minute in three minute intervals increased to 20, 30, 40 or 50 micrograms/kg per minute or to a peak heart rate response of at least 85% age predicted maximum heart rate. If at the end of the Dobutamine protocol, there is inadequate heart rate response, intravenous atropine boluses of 0.5 milligrams (maximum 1.0 mg) would be used as needed to achieve a heart rate of at least 85% of age predicted maximum heart rate.
Period: Overall Study
Arm/Group | Dobutamine Stress Echo (DSE)
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dobutamine Stress Echo (DSE)
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricle Mean Diastolic Pressure
Description: Left ventricle filling pressures were measured using a pigtail catheter inserted into the left ventricle. Measurements of left ventricle pressures were taken at baseline, 3 minutes, 6 minutes, 9 minutes, 12 minutes, and recovery. Change from baseline at recovery reported.
Time Frame: Baseline, recovery
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Dobutamine Stress Echo (DSE)
Number analyzed (Participants) | 16
mmHg | 3.3 [3.0 to 3.6]

2. Secondary Outcome: Change in Early Transmitral Velocity/Early Lateral Mitral Velocity (E/E')
Description: Echocardiography was performed at rest and with dobutamine stress at 3 minutes, 6 minutes, 9 minutes, and 12 minutes, to measure differences in E/E' at the septum and lateral mitral annulus. Change from baseline at recovery reported.
Time Frame: Baseline, recovery
Measure: Mean (Full Range); unit: Ratio
Arm/Group | Dobutamine Stress Echo (DSE)
Number analyzed (Participants) | 16
Ratio
  Septum E/E' | 0.4 [-1.3 to 0.5]
  Lateral E/E' | -0.4 [-2 to 1.2]

ADVERSE EVENTS:
Arm/Group | Dobutamine Stress Echo (DSE)
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes